CLINICAL TRIAL: NCT00335777
Title: An Open-Label Pilot Trial To Collect And Evaluate Data On The Use Of Migranal® In The Treatment Of Two Acute Migraine Attacks Associated With Cutaneous Allodynia
Brief Title: A Research Study Examining Migranal and Skin Sensitivity in Subjects With Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SDS/MIG-CA/ 01
Record Dates: First submitted 2006-06-09; First posted 2006-06-12 (Estimated); Results first posted 2011-10-14 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Dihydroergotamine

ARMS (2):
- Migranal treatment first treatment phase (Experimental): All subjects were asked to treat one headache at 1 hour (early) and one headache at 4 hours after onset of throbbing (late). Dose of nasal spray constant for both time points. The subject could determine the order in which they could treat the headaches (early (first treatment phase) then late (second treatment phase), or late (first treatment phase) then early (second treatment phase).
  Interventions: Drug: Migranal nasal spray at 1 hour
- Migranal second treatment phase (Experimental): All subjects were asked to treat one headache at 1 hour (early) and one headache at 4 hours after onset of throbbing (late). Dose of nasal spray constant for both time points. The subject could determine the order in which they could treat the headaches (early (first treatment phase) then late (second treatment phase), or late (first treatment phase) then early (second treatment phase).
  Interventions: Drug: Migranal nasal spray at 4 hour

INTERVENTIONS:
Drug: Migranal nasal spray at 1 hour — Migranal® 4 mg. will be self administered by each subject in the following manner: one spray in each nostril, wait 15 minutes then follow with one spray in each nostril. This will deliver the desired 4 mg. dose.
  Other Names: Dihydroergotamine (DHE)
  Arms: Migranal treatment first treatment phase
Drug: Migranal nasal spray at 4 hour — Migranal® 4 mg. will be self administered by each subject in the following manner: one spray in each nostril, wait 15 minutes then follow with one spray in each nostril. This will deliver the desired 4 mg. dose.
  Other Names: Dihydroergotamine (DHE)
  Arms: Migranal second treatment phase

SUMMARY:
This is a research study looking at Migranal (study drug) in the treatment of two migraine attacks in patients who have a history of cutaneous allodynia (pronounced q-tay-nee-us al-o-din-ee-a). Cutaneous allodynia is an increased skin sensitivity experienced during a headache. It has been noted in several studies that in patients with migraine, seventy nine percent of the patients experienced allodynia on the facial skin on the same side as the headache. Understanding more about allodynia may help us understand how the pain system works in migraine.

This study will compare the differences, if any, in attacks treated early with study drug (at 1-hour from onset) and attacks treated later (at 4-hours). You will be asked to treat one attack early and one attack late for this study. If the first attack you treat is early (at 1 hour following onset of throbbing pain) then the second attack you treat should be late (at 4 hours following onset of throbbing pain).

It is hoped that this study will provide information on the use of Migranal in subjects who have cutaneous allodynia. The results from this study may be used in the development of larger clinical trials. The study drug is a medication that is taken in the form of nasal spray.

DETAILED DESCRIPTION:
This is a three visit trial consisting of a screening visit, one follow-up visit and a termination visit. Subjects will be screened using the Cutaneous Allodynia Screening Tool (Appendix A) and the investigator will determine whether or not the subject experiences episodic migraine headaches associated with cutaneous allodynia. Those subjects who test positive for the afore-stated will then proceed with the treatment phase of the project.

Migranal® will be taken by the subject at home at 1-hour following the onset of throbbing pain for one of the two qualifying migraine attacks and at 4-hours following onset of throbbing pain for the second qualifying migraine attack. Migranal® 4 mg. will be self administered by each subject in the following manner: one spray in each nostril, wait 15 minutes then follow with one spray in each nostril. This will deliver the desired 4 mg. dose. Cutaneous allodynia assessments will be made periodically prior to and after administration of study drug. Subjects will be asked to return to the center within 1 week of treating each attack. Subjects will be instructed to treat their 1st qualifying attack within 6 weeks of the screening visit and their 2nd qualifying attack within 6 weeks of their follow-up visit 1.

Migraine pain and associated symptoms assessments will be measured by the subjects for 24-hours from the administration of study drug for each attack.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the ages of 18 and 65, inclusive
* Subjects diagnosed with episodic migraine, with or without aura according to IHS (International Headache Society) criteria (Appendix B) for at least one-year prior to screening
* Subjects who experience between 3-10 migraine attacks (inclusive) per month (during the previous 6 months) with no more than 15 days of headache per month.
* Subjects who report their migraine pain quality as pulsating/ throbbing.
* Subject experiences episodic migraine associated with cutaneous allodynia, as determined by the Cutaneous Allodynia screening tool and investigator.
* Subject is using or agrees to use for the duration of participation a medically acceptable form of contraception (as determined by investigator), if female of child-bearing potential
* Subjects who are able to understand and comply with all study procedures.
* Subject provides written informed consent prior to any screening procedures being conducted

Exclusion Criteria:

* Pregnant and/or lactating women
* Subjects who, in the investigators opinion, have a history or have evidence of a medical or psychiatric condition that would expose them to an increased risk of a significant adverse event or would interfere with the assessments of efficacy and tolerability during this trial
* Subjects with an abnormal ECG that, in the investigators opinion, would expose them to increased risk of adverse events or interfere with study drug and/or analysis of efficacy/tolerability
* Subjects currently using, or expecting to use during the trial, CYP 3A4(CYP3A4 enzyme) inhibitors (such as protease inhibitors and macrolide antibiotics)
* Subjects with severely impaired hepatic or renal function, as determined by the investigator
* Subjects who have participated in an investigational drug trial in the 30 days prior to the screening visit
* Subjects who currently have or have a history of basilar or hemiplegic migraine
* Subjects who have previously shown hypersensitivity to ergot alkaloids
* Subjects who have a history of non-response to DHE-45 (dihydroergotamine) or Migranal®, as determined by investigator
* Subjects with uncontrolled hypertension
* Subjects who currently have or who have a history of ischemia and/or vasospastic coronary artery disease
* Subjects who, in the investigators opinion, have significant risk factors of coronary artery disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2006-08; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D. Silberstein, M.D., Principal Investigator — Jefferson Headache Center
Locations (1):
- Jefferson Headache Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from our office practice or surrounding community and screened at the Jefferson Headache Center between 8/21/06 and 6/18/08.
Pre-assignment Details: Eligible subjects were enrolled in the study and dispensed open label study medication at the end of the screening visit.
Groups:
- Migranal: All Subjects: All subjects enrolled in study
Period: Enrolled and Dispensed Study Medication
Arm/Group | Migranal: All Subjects
Started | 64 (64 subjects enrolled. 35 treated 2 headaches, but 22/35 at appropriate times, as per protocol.)
Completed | 35
Not Completed | 29
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 6
Not completed — Treated only 1 or no headaches | 18
Period: Treated 2 Headaches Per Protocol
Arm/Group | Migranal: All Subjects
Started | 35
Completed | 22
Not Completed | 13
Not completed — Treated 2 early or 2 late headaches | 1
Not completed — Treated out of protocol for early and late | 12

BASELINE CHARACTERISTICS:
Arm/Group | Migranal: All Subjects
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.86 (10.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 64

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Were Pain Free at 2 Hours Post Treatment With Study Drug.
Description: Number of subjects who were pain free at 2 hours after treatment with study medication when they treated a migraine early (defined as treatment within 1 hour of onset of throbbing pain) compared to the number of subjects who were pain free at 2 hours after treatment with study medication when they treated late (defined as 4 hours after onset of throbbing pain). "Pain free" is defined as a subject rating of zero on a 4 point pain scale; (0=None, 1=mild, 2= moderate, 3=severe).
Time Frame: 2 hours post treatment with study medication
Population: Per protocol population was used in the efficacy analyses. 22 subjects were included, since they treated a migraine early and another migraine late, as defined in the protocol, with study medication.(Cross-over design)
Measure: Number; unit: participants
Groups:
- Migranal: Early Treatment: Treated headache within 1.25 hours of onset of throbbing
- Migranal Late Treatment: Treated a headache at greater or equal to 3.5 hours after onset of throbbing
Arm/Group | Migranal: Early Treatment | Migranal Late Treatment
Number analyzed (Participants) | 22 | 22
participants | 4 | 8
Statistical Analysis 1: Comparison: Migranal: Early Treatment vs Migranal Late Treatment; Null hypothesis: there is no difference in the proportion of subjects who were pain free when treating early, as compared to treating late; Test type: Non-Inferiority or Equivalence — 2 sided McNemar test; p = 0.289, McNemar; 2 sided McNemar

2. Secondary Outcome: Number of Subjects Who Had Pain Relief at 2 Hours Post Treatment With Study Drug.
Description: Number of subjects who had pain relief at 2 hours after treatment with study medication when they treated a migraine early (defined as treatment within 1 hour of onset of throbbing pain) compared to the number of subjects who were pain relief at 2 hours after treatment with study medication when they treated late (defined as 4 hours after onset of throbbing pain). "Pain reduction" is defined as a subject with a 1 or more point decrease on a 4 point pain scale; (0=None, 1=mild, 2= moderate, 3=severe).
Time Frame: 2 hours post treatment with study medication
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Migranal: Early Treatment | Migranal Late Treatment
Number analyzed (Participants) | 22 | 22
Participants | 14 | 15
Statistical Analysis 1: Comparison: Migranal: Early Treatment vs Migranal Late Treatment; Null hypothesis: there is no difference in the proportion of subjects who had pain relief when treating early, as compared to treating late; Test type: Non-Inferiority or Equivalence — 2 sided McNemar test; p = 1.000, McNemar; 2 sided McNemar test

ADVERSE EVENTS:
Time Frame: Adverse Events collected from time of dosing through 48 hours post dose.
Description: Adverse Event assessments were performed on all subjects who took any study medication, even if they did not treat according to the guidelines in the protocol. N=48
Arm/Group | Migranal: All Subjects
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 14/48
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Migranal: All Subjects (N=48)
mouth and throat discomfort (General disorders) | 3
nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 5 — nasal burning, stuffiness or discomfort
nausea (Gastrointestinal disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes